CLINICAL TRIAL: NCT01639287
Title: Correlation of "Painless" Synovitis With Clinical, Laboratory and Radiological (X-ray, Sonography) Finds in Patients With Longstanding Rheumatoid Arthritis (RA).
Brief Title: Painless Synovitis in Patients With Longstanding Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Daniele Freitas Pereira, Dr, Principal Investigator, Federal University of São Paulo
Other Study IDs: USG-3131-AR
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: - Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Painless: Painless synovitis group(called "cold" synovitis)
- Painful: Painful synovitis group

SUMMARY:
There is a group of patients with rheumatoid arthritis (RA) that suffer from chronically painless synovitis in the hands.

The objective of this study is to compare painless synovitis with painful synovitis according to the sonographic (Gray-scale and power Doppler) findings.

A sonographic examination (Gray-scale and power Doppler) will be done to evaluate metacarpophalangeal joints of patients without local painful and will be a comparison with patients with local painful.

DETAILED DESCRIPTION:
Introduction/Objectives:

There is a group of patients with rheumatoid arthritis (RA) that suffer from chronically painless synovitis in the hands. The mean of this is still unknown and does not exist studies in the literature that assessing the predictors of this behavior or synovial potential to cause bone erosion.

The objective of this study is to compare painless synovitis (called "cold" synovitis) with painful synovitis according to the sonographic (Gray-scale and power Doppler) findings, articular damage (x-Ray and sonography), clinical, laboratory and demographic variables in RA patients.

Methods: Cross-sectional study with RA patients, which will be evaluated metacarpophalangeal joints of patients without local painful. Sixty RA patients will be selected in the Federal University of São Paulo ambulatory (Unifesp). The patients will be divided in two groups of thirty patients each: "painless synovitis" Group and "painful synovitis" Group. All patients will be measured through clinical evaluation, hands ultrasound and laboratory parameters (erythrocyte sedimentation rate, ESR; rheumatoid factor, RF; anti-cyclic-citrullinated peptide antibodies, CCP) on the same day. The clinical evaluation will be measured by a trained rheumatologist with experience in joint physical examination (synovitis). This measure will be done before the sonography examination and the assessment tools will be: painful joint count; swollen joint count; painful visual analogue scale (VAS 0-10); swollen VAS; activity disease VAS; measurement of grip strength and pinch with Jamar dynamometer and Preston Pinch Gauge; 28 joint Disease Activity Score (DAS 28); Stanford Health Assessment Questionnaire (HAQ); Cochin Hand Functional Scale (CHFS) and patient clinical evaluation. The level of statistical significance will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* longstanding rheumatoid arthritis
* chronically painless synovitis in the hands or painful

Exclusion Criteria:

* uncompensated systemic disease, e.g. diabetes mellitus, hypothyroidism
* change of basic drug in the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Federal University of São Paulo ambulatory (Unifesp) and basic helth unit
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Sonographic power Doppler | baseline

SECONDARY OUTCOMES:
Sonographic Gray Scale | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Daniele F Pereira, Dr, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil